CLINICAL TRIAL: NCT03235037
Title: Clinical Trial of Levodopa/Carbidopa ( Sinemet) Therapy in Angel Man Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bennett Lavenstein (Other)
Responsible Party: Sponsor-Investigator, Bennett Lavenstein, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB PRO00004116
Record Dates: First submitted 2017-07-28; First posted 2017-08-01 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Angelman Syndrome
MeSH Terms: conditions — Angelman Syndrome | interventions — Levodopa; carbidopa, levodopa drug combination

STUDY DESIGN:
Intervention Model Description: This is an open label study to assess the motor and cognitive and developmental effects of carbidopa/levodopa when administered orally in doses of 1 -10mg per kg per day. This study will recruit and monitor patients over a 2 year period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sinemet (Other): The target dose of Sinemet is 2-10 mg per kilogram per day of levodopa. The initial dose will be determined by your weight and age and will start at a low dosage level, 1 mg per kilogram per day. The dose will be re-evaluated after the first 2 weeks and may be adjusted at each visit depending on your response to the drug.
  Interventions: Drug: Levodopa

INTERVENTIONS:
Drug: Levodopa — The target dose of Sinemet is 2-10 mg per kilogram per day of levodopa. The initial dose will be determined by your weight and age and will start at a low dosage level, 1 mg per kilogram per day. The dose will be re-evaluated after the first 2 weeks and may be adjusted at each visit depending on your response to the drug.
  Other Names: Sinemet

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness (how well a drug works) of Carbidopa/levodopa (Sinemet) in individuals with Angelman syndrome. Sinemet is a medication that helps to raise dopamine levels (a chemical that signals nerve cells) in the brain and central nervous system. There is evidence that dopamine concentrations may be abnormal in patients with Angelman syndrome. This study is investigating whether Sinemet helps motor control, intellectual function and the achievement of developmental milestones in people with Angelman syndrome

DETAILED DESCRIPTION:
Angelman syndrome (AS) is a well-recognized cause of disability in children who present with movement or balance disorder, usually ataxia and/or tremulous movement of the limbs, severe speech and cognitive delay behavior disorders and was initially described by Harry Angelman as the " happy puppet syndrome" due to their disposition. Seizures, abnormal sleep-wake cycles and distinctive facial features have been also commonly seen. This disorder is almost exclusively diagnosed in childhood but adults have been reported. Angelman syndrome affects an estimated 1 in 12,000 to 20,000 people. Many of the characteristic features are caused by the loss of function of maternally inherited UBE3A allele on chromosome 15q11-q13 locus. Several different genetic mechanisms can cause loss of function of maternally inherited UBE3A gene. Majority of AS is caused by deletion of chromosome 15q11.2-q13 (approximately 70%), 11% is caused by a mutation in maternal copy of UBE3A. Paternal uniparental disomy (pat UPD) occurs in 7%. Rarely, a defect in imprinting region and chromosome rearrangement can also lead to AS.

Ubiquitin-protein ligase E3A (UBE3A) is involved in protein degradation through the ubiquitin proteasome pathway and displays predominantly in human fetal brain and adult frontal cortex. UBE3a is essential in the regulation of GTP cyclohydrolase I, an essential enzyme in dopamine biosynthesis. Knockout mouse studies have evaluated dopamine dependent behaviors as well as dopamine synthesis, content and release in the mesolimbic and nigrostriatal pathway of AS model mice. Impairment of UBE3A results in the accumulation of protein substrate and is also associated with a loss of dopaminergic neuronal function which plays a role in the clinical symptomatology. AS ( knockout) mice were reported to have maternal deficiency of Ube3a with reduced dopamine cell number in the substantia nigra pars compacta ((basal ganglia) . They demonstrated motoric and cognitive deficits. There are several mouse models that have demonstrated both the disorder and the beneficial effect of L dopa in the knockout mouse providing a basis for clinical human trials.

To date the primary treatment of children with Angelman syndrome has been only supportive and symptomatic such as physical, occupation and speech therapies, melatonin and Benadryl for insomnia and the treatment of seizure disorders. Little attention or success has been directed to the primary gait disturbance, namely ataxia and the cognitive impairment including processing, attention and speech delays which are cardinal features of the disorder.

In 2001, Harbord has reported two adults with Angelman syndrome and Parkinson's disease who had a positive response to L Dopa constituting the first report of the use of levodopa in Angelman syndrome.

Pediatric neurotransmitter disorders have previously been recognized involving the dopamine pathway. In the past investigators have reported on the distinct developmental and behavioral profile, cognitive deficits, motor and language skills utilizing standardized testing in the NIH Rare Disease Clinical Research Network, Angelman Rett collaborative.

This study will look at the effects of L Dopa on motor control including ataxia, cognitive function and developmental milestones in subjects with Angelman syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Angelman syndrome confirmed by molecular genetic testing.
* Age between 18 months and 16 years of age
* Absence of any contraindication to the use of Sinemet as determined by the PI

Exclusion Criteria:

* Intractable epilepsy not responsive to anticonvulsive therapy in the patient with this syndrome.
* History of prior drug intolerances/drug hypersensitivity to any agent that may be similar to L Dopa .
* Progressively deteriorating EEG pattern.

Ages: 18 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2013-11-26 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Improvement in motor control determined through composite measure- Tremor | 2 years
  Documented improvement in motor control including tremor using SARA Scale ( Short Ataxia Rating Assesment)
Improvement in motor control determined through composite measure-Ataxia | 2 years
  Documented improvement in motor control including ataxia, using SARA Scale ( Short Ataxia Rating Assesment)
Improvement in motor control determined through composite measure- SARA score | 2 years
  Documented improvement in SARA score

SECONDARY OUTCOMES:
Improvement in development determined through composite measure-Psychoeducational Testing | 2 years
  Documented improvement in development based upon Bailey, Denver, Vanderbilt, Educational testing.

CONTACTS AND LOCATIONS:
Overall Officials: Bennett Lavenstein, MD, Principal Investigator — Children's National Health System, Department of Neurology